CLINICAL TRIAL: NCT06994234
Title: Effect of In-Place Slow Jogging on Metabolic Dysfunction-Associated Steatotic Liver Disease: A Prospective Randomized Controlled Trial
Brief Title: Effect of In-Place Slow Jogging on Metabolic Dysfunction-Associated Steatotic Liver Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025YS-079
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Metabolic Dysfunction-Associated Steatotic Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-Place Slow Jogging Group (Experimental): During the 3-month intervention period, the diet followed the outpatient health prescription of MASLD, and ultra-jogging training was carried out 5 times a week, and each training session lasted for 30 minutes.
  Interventions: Behavioral: In-Place Slow Jogging
- Control Group (No Intervention): During the 3-month intervention period, the diet followed the health prescription of our MASLD outpatient clinic, and patients were encouraged to maintain their daily physical activity level, such as walking up and down stairs, walking short distances, etc. However, there is no in-situ ultra-jogging intervention.

INTERVENTIONS:
Behavioral: In-Place Slow Jogging — ultra-jogging training was carried out 5 times a week, and each training session lasted for 30 minutes.
  Arms: In-Place Slow Jogging Group

SUMMARY:
Evaluating the Effectiveness, Safety, and Feasibility of Stationary Ultra-Slow Running in Treating MASLD Patients.

ELIGIBILITY:
Inclusion Criteria:

1. Meeting the diagnostic criteria for MASLD.
2. Aged between 18 and 70 years (inclusive), regardless of gender.
3. Patients voluntarily participate in this clinical study, have signed the informed consent form, and agree to comply with all study requirements, including follow-up visits, examinations, and treatments.

Exclusion Criteria:

1. Exclusion of other conditions causing liver injury, including alcoholic hepatitis, active hepatitis B or C virus infection, drug-induced hepatitis, autoimmune hepatitis, primary sclerosing cholangitis, Wilson's disease, α1-antitrypsin deficiency, liver cancer (or family history of liver cancer), etc.
2. History of medication use for more than 2 weeks within the past year that may induce hepatic steatosis or steatohepatitis (e.g., amiodarone, methotrexate, systemic glucocorticoids, tetracycline, tamoxifen, estrogen exceeding hormone replacement doses, anabolic steroids, valproic acid, or other known hepatotoxins).
3. Use of hepatoprotective drugs (including but not limited to reduced glutathione, glucurolactone, glycyrrhizin preparations, nicotinamide, bifendate, liver-protecting tablets, silymarin, polyene phosphatidylcholine, S-adenosylmethionine, ursodeoxycholic acid, vitamin E, or other herbal medicines affecting liver function) within 4 weeks prior to enrollment.
4. Presence of ascites, variceal bleeding, hepatic encephalopathy, spontaneous bacterial peritonitis, or history of liver transplantation at randomization or previously, or planned liver transplantation.
5. Concurrent type 1 diabetes.
6. Severe cardiovascular, cerebrovascular, renal, or hematopoietic system diseases, as well as mood disorders (e.g., anxiety, depression) or psychiatric illnesses.
7. Patients with any type of malignancy or a history of malignancy.
8. HIV-positive status.
9. Pregnant or breastfeeding women, or subjects of childbearing potential unwilling or unable to use effective contraception from the screening period until 6 months after discontinuation of the investigational drug.
10. Participation in other interventional clinical trials within 12 weeks prior to screening.
11. Patients with unstable weight (i.e., weight loss or gain exceeding 4 kg in the past 3 months) or those with conditions preventing participation in the exercise program.
12. Other conditions deemed by the investigator as unsuitable for participation in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2025-06-20 (Estimated); Primary Completion 2027-06-20 (Estimated); Study Completion 2028-06-20 (Estimated)

PRIMARY OUTCOMES:
Liver Stiffness Measurement (LSM) | Baseline, 3 months post-treatment
  Measure method：FibroScan
Controlled Attenuation Parameter(CAP) | Baseline, 3 months post-treatment
  Measure method：FibroScan

SECONDARY OUTCOMES:
Polysomnography metrics | Baseline, 3 months post-treatment
  Measure method:Polysomnography（PSG)
Height | Baseline, 1 months post-treatment, 2 months post-treatment, 3 months post-treatment
Body Weight | Baseline, 1 months post-treatment, 2 months post-treatment, 3 months post-treatment
Waist Circumference | Baseline, 1 months post-treatment, 2 months post-treatment, 3 months post-treatment
Body Fat Percentage | Baseline, 1 months post-treatment, 2 months post-treatment, 3 months post-treatment
Lean Body Mass | Baseline, 1 months post-treatment, 2 months post-treatment, 3 months post-treatment
BMI | Baseline, 1 months post-treatment, 2 months post-treatment, 3 months post-treatment
albumin | Baseline, 1 months post-treatment, 2 months post-treatment, 3 months post-treatment
  The unit is grams per liter (g/L). It reflects liver synthetic function and nutritional status. Normal reference values are 35-50 g/L for adults and 34-48 g/L for individuals aged 60 years or older.Time
Hemoglobin | Baseline, 1 months post-treatment, 2 months post-treatment, 3 months post-treatment
  The unit is grams per liter (g/L). It is used to assess anemia or polycythemia. Normal reference values are as follows: adult males: 120-160 g/L; adult females: 110-150
body temperature | Baseline, 1 months post-treatment, 2 months post-treatment, 3 months post-treatment
  The unit is degrees Celsius (℃). Normal range: axillary temperature is 36℃ to 37℃.Time Frame: Baseline, at 1 week, 4 weeks, 8 weeks, and 12 weeks after
Respiratory Rate | Baseline, 1 months post-treatment, 2 months post-treatment, 3 months post-treatment
  The unit is breaths per minute (breaths/min). Normal range: adults, 16-20 breaths/min (at rest).Tachypnea may be caused by reasons such as pneumonia, fever, cardiovascular diseases, anemia, etc., while bradypnea may be caused by reasons such as increased intracranial pressure, hypothyroidism, etc.
Blood Pressure | Baseline, 1 months post-treatment, 2 months post-treatment, 3 months post-treatment
  The unit is millimeters of mercury (mmHg). Normal range: systolic pressure, 90-139 mmHg; diastolic pressure, 60-89 mmHg.
Heart Rate | Baseline, 1 months post-treatment, 2 months post-treatment, 3 months post-treatment
  The unit is beats per minute (beats/min). Normal range: 60-100 beats/min (at rest).
Blood White Blood Cells | Baseline, 1 months post-treatment, 2 months post-treatment, 3 months post-treatment
  Normal range for adults is 4.0-10.0×10⁹/L. An elevated level may indicate bacterial infection or inflammation, while a decreased level may be associated with viral infections or drug reactions.
Bloos Red Blood Cells | Baseline, 1 months post-treatment, 2 months post-treatment, 3 months post-treatment
  Normal range is 4.3-5.8×10¹²/L for males and 3.8-5.1×10¹²/L for females.
Platelets | Baseline, 1 months post-treatment, 2 months post-treatment, 3 months post-treatment
  Normal range is 125-350×10⁹/L. A reduced count increases the risk of bleeding, while an elevated count increases the risk of thrombosis.
alanine aminotransferase (ALT) | Baseline, 1 months post-treatment, 2 months post-treatment, 3 months post-treatment
  Normal range is 7-40 U/L. Elevated levels indicate liver damage.Time
aspartate aminotransferase (AST) | Baseline, 1 months post-treatment, 2 months post-treatment, 3 months post-treatment
  Normal range is 13-35 U/L. Elevated levels indicate liver damage.
serum creatinine (Cr) | Baseline, 1 months post-treatment, 2 months post-treatment, 3 months post-treatment
  Normal range is 53-106 μmol/L for males and 44-97 μmol/L for females. Elevated levels suggest decreased renal function.
Blood Urea Nitrogen (BUN) | Baseline, 1 months post-treatment, 2 months post-treatment, 3 months post-treatment
  Normal range is 2.9-7.5 mmol/L. Elevated levels may be associated with renal failure or dehydration.
Total Cholesterol (TC) | Baseline, 1 months post-treatment, 2 months post-treatment, 3 months post-treatment
Triglycerides (TG) | Baseline, 1 months post-treatment, 2 months post-treatment, 3 months post-treatment
High-Density Lipoprotein Cholesterol（HDL) | Baseline, 1 months post-treatment, 2 months post-treatment, 3 months post-treatment
Fasting Blood Glucose (FBG) | Baseline, 1 months post-treatment, 2 months post-treatment, 3 months post-treatment
Fasting Insulin (FINS) | Baseline, 1 months post-treatment, 2 months post-treatment, 3 months post-treatment
Hyaluronic Acid（HA) | Baseline, 1 months post-treatment, 2 months post-treatment, 3 months post-treatment
Procollagen III N-Terminal Peptide（PIIINP) | Baseline, 1 months post-treatment, 2 months post-treatment, 3 months post-treatment
Collagen Type IV（CIV) | Baseline, 1 months post-treatment, 2 months post-treatment, 3 months post-treatment
Laminin（LN) | Baseline, 1 months post-treatment, 2 months post-treatment, 3 months post-treatment
Glycated Hemoglobin (HbA1c) | Baseline, 1 months post-treatment, 2 months post-treatment, 3 months post-treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No